CLINICAL TRIAL: NCT02398240
Title: A Pilot Study of Risk Adapted Therapy Utilizing Upfront Brentuximab With Combination Chemotherapy in the Treatment of Children, Adolescents and Young Adults With Newly Diagnosed Hodgkin Lymphoma
Brief Title: Brentuximab for Newly Diagnosed Hodgkin Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mitchell Cairo (Other)
Responsible Party: Sponsor-Investigator, Mitchell Cairo, Executive Vice Chair, New York Medical College
Organization: New York Medical College (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-568
Record Dates: First submitted 2015-03-15; First posted 2015-03-25 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Doxorubicin; liposomal doxorubicin; Vincristine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Risk (Experimental): Low Risk Patients (Stage IA, IIA; no bulky disease or extension): 3 cycles of chemotherapy
  Interventions: Drug: Brentuximab Vedotin; Drug: Doxorubicin; Drug: Vincristine
- Intermediate Risk (Experimental): Intermediate Risk Patients (Stage IA bulk/E, IB, IIA bulk/E, IIB, IIIA): 4 cycles of chemotherapy
  Interventions: Drug: Brentuximab Vedotin; Drug: Doxorubicin; Drug: Vincristine; Drug: Rituximab
- High Risk (Experimental): High Risk Patients (Stage IIIA bulk/ E, IIIB, IVA/B): 6 cycles of chemotherapy
  Interventions: Drug: Brentuximab Vedotin; Drug: Doxorubicin; Drug: Vincristine; Drug: Rituximab

INTERVENTIONS:
Drug: Brentuximab Vedotin — Day 1 and 15 Dose: 1.2 mg/kg/dose. (Maximum dose is 120 mg)
  Other Names: Adcetris
Drug: Doxorubicin — Days: 1 and 15 Dose: 25 mg/m2/dose.
  Other Names: Doxil, Adriamycin
Drug: Vincristine — Days: 1 and 15 Dose: 1.5 mg/m2/dose (max: 2 mg/dose).
  Other Names: Oncovin
Drug: Rituximab — Days: 2 and 16 Dose: 375 mg/m2/dose.
  Other Names: Rituxan
  Arms: High Risk; Intermediate Risk

SUMMARY:
The addition of Brentuximab vedotin (Bv) to combination chemotherapy will be safe, well tolerated and effective in children, adolescents and young adults with all stages of newly diagnosed Hodgkin lymphoma (HL).

ELIGIBILITY:
Inclusion Criteria:

* Normal Serum creatinine based on age or creatinine clearance >60 ml/min/1.73 m2 or an equivalent radioisotope glomerular filtration rate (GFR) as determined by the institutional normal range.
* Direct bilirubin < 1.5 upper limit of normal (ULN) for age, and SGOT (AST) or SGPT (ALT) <3 x ULN
* Shortening fraction >27% by echocardiogram, or
* Ejection fraction of >50% by radionuclide angiogram or echocardiogram.
* For patients age 1-16 years, Lansky score of ≥60.
* For patients > 16 years, Karnofsky score of ≥60.
* No prior Hodgkin lymphoma directed therapy is allowed except for emergent mediastinal irradiation (<1000cGy) for superior vena cava (SVC) syndrome.

Exclusion Criteria:

* Females who are pregnant (positive HCG) or lactating.
* Karnofsky <60% or Lansky <60% if less than 16 years of age.
* Age ≤1 year or >29.99 years of age.

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
To determine if this combination of chemoimmunotherapy is safe to administer. (Adverse events) | 1 year
  Adverse events will be monitored each cycle to determine if there are any events related possibly, probably or definitely related to study therapy
To determine the response rate | 1 year
  disease evaluations will be performed after the 2nd, 4th and 6th cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Hochberg, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hochberg J, Basso J, Shi Q, Klejmont L, Flower A, Bortfeld K, Harrison L, van de Ven C, Moorthy C, Islam H, Gerard P, Voss S, Cairo MS. Risk-adapted chemoimmunotherapy using brentuximab vedotin and rituximab in children, adolescents, and young adults with newly diagnosed Hodgkin's lymphoma: a phase II, non-randomized controlled trial. J Immunother Cancer. 2022 May;10(5):e004445. doi: 10.1136/jitc-2021-004445. PMID 35584865